CLINICAL TRIAL: NCT04790058
Title: Implementation of Canadian Syncope Risk Score Based Practice Recommendations for Emergency Department Syncope Management - A Pilot Study
Brief Title: CSRS Implementation - A Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Queensway Carleton Hospital (Other)
Responsible Party: Principal Investigator, Venkatesh Thiruganasambandamoorthy, Principal Investigator, Ottawa Hospital Research Institute
Other Study IDs: CRF 2589
Record Dates: First submitted 2020-12-11; First posted 2021-03-10 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Syncope
Keywords: Syncope; Emergency Department; Risk Stratification
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Physicians using CSRS practice recommendation to treat syncope patients in ED.: During the control period, there will be no interventions. The intervention is the knowledge translation of the CSRS practice recommendations. The components of the practice recommendations include: 1) evidence-informed systematic clinical evaluation with appropriate history, physical examination and in-ED investigations (e.g. troponin testing, work-up for pulmonary embolism and CT head) for detecting serious underlying conditions and predicting 30-day serious outcomes; 2) application of the CSRS for risk-stratification at the end of ED visit after no serious underlying conditions for the syncope were identified; 3) use of patient information materials to aid in disposition; 4) the use of 15-day outpatient cardiac monitoring for CSRS medium and high-risk patients upon ED discharge. The ED physician or non-ED physician performing consultation on the patient can apply all the components of the practice recommendation and decide disposition of the patients who are eligible to be studied.
  Interventions: Other: Knowledge translation of the CSRS practice recommendations

INTERVENTIONS:
Other: Knowledge translation of the CSRS practice recommendations — The intervention is knowledge translation of the CSRS practice recommendations; the application of the practice recommendations will occur during the patient's ED visit and patients who are eligible for 15-day cardiac rhythm monitoring will have Holter monitor applied at the time of ED discharge. For the secondary objective to validate the accuracy of the ultra-low risk criteria of CSRS and assess for potential improvements in the practice recommendations and the prediction models we will request verbal consent during the index ED visit for addition of cardiac biomarker measurements [troponin and NT-proBNP] for patients who did not have such measurements performed as part of routine clinical care, and a 30-day telephone follow-up for serious outcome assessment. Patients who do not consent will be excluded from these portions of the study but included in the health resource utilization and generic patient safety outcome assessment objectives.

SUMMARY:
Syncope is a common reason for emergency department (ED) presentation. While often benign, some patients have serious and life-threatening underlying causes, both cardiac and non-cardiac, which may or may not be apparent at the time of the initial ED assessment. Identifying which patients will benefit from further investigation, ongoing monitoring and/or hospital admission is essential to reduce both adverse outcomes and the high costs. Our group has spent over a decade developing the evidence base for a risk stratification tool directed at optimizing the accuracy of ED decisions: the Canadian Syncope Risk Score (CSRS). This tool is now ready for the final phase of its introduction into clinical practice, namely a robust, multicentre implementation trial of the CSRS based practice recommendations to demonstrate its real-world effectiveness. Prior to the launch of the large-scale implementation trial, a pilot study to assess primarily the feasibility and secondarily the effectiveness is needed.

DETAILED DESCRIPTION:
ED crowding limits the ability of the emergency providers to provide quality care, is a growing crisis in North America and Europe, and leads to unsafe and rushed disposition decisions which compromise patient care. On the other hand, hospital admission is expensive, and an increasing awareness of nosocomial morbidity and the harms of unnecessary testing and hospitalization exert countervailing pressure on low-yield admissions from the ED. Therefore, improved accuracy in ED disposition decision-making is more important than ever, and syncope typifies a common, high stakes condition in which improvements in efficiency are badly needed.

Identifying which patients will benefit from further cardiac rhythm monitoring and/or hospital admission is essential to reduce both adverse outcomes and high costs. A comprehensive literature review of risk-tools and international guidelines concede that previously published tools lack or have failed external validation, are excessively complex, include as outcomes obvious conditions readily identified during the index ED evaluation, or lacked power and specificity. These tools also do not offer specific clinical actions and are not supported by the guidelines. The CSRS addresses each of the above weaknesses and coupled with outpatient live cardiac monitoring is an innovative and standardized approach to ED syncope management to expedite ED care, improve patient safety and reduce healthcare costs. The investigators have identified the barriers and facilitators to effectively adapt knowledge into local contexts as per the Knowledge to Action cycle, and have selected implementation strategies accordingly. The proposed pilot study is a right step before widescale implementation.

The primary objective of this pilot study is to assess the feasibility of implementing the practice recommendations. The secondary objectives are to assess the effectiveness and safety of the intervention, implementation of the CSRS-based practice recommendations. Specific objectives include:

Feasibility objectives:

Primary: to assess the reach of the intervention Secondary: to assess the adoption, adherence, and sustainability of the intervention; to assess the acceptability, the feasibility of use and the complexity of the intervention; and to assess the satisfaction to the dose (i.e., exposure) of the intervention received including support and resources.

Effectiveness objectives:

Primary: to assess the impact on ED disposition time, defined as the time interval between ED physician initial assessment and ED disposition.

Secondary: to assess the impact on hospitalizations, investigations and consultations performed in the ED.

Safety objective: To assess mortality, return ED visits and hospitalization within 30-days and 1-year of the index ED visit (generic patient safety outcome) and to monitor the safety of the CSRS application by assessing the 30-day serious outcomes after ED disposition (syncope specific short-term serious outcome).

We will conduct the study over a 9-month period, with the TOH and QCH EDs receiving the intervention at the 3rd and 4th month respectively. The first month of the intervention period will be designated as a transition period during which we will undertake intense educational efforts. The total intervention period for the QCH and TOH EDs will be 5 and 6 months respectively.

ELIGIBILITY:
1. Physician: physicians involved in ED syncope care
2. Patients:

   * Inclusion Criteria: adult (aged > 18 years) patients who present within 24 hours of syncope
   * Exclusion Criteria:

     * non-syncope (prolonged LOC >5 minutes, change in the mental status from baseline, patients with witnessed obvious seizure, or head trauma preceding the LOC),
     * those unable to provide proper details - e.g., intoxication, and those with significant trauma requiring admission as per international consensus.
     * patients who had a serious underlying condition identified during the index ED evaluation
     * hospitalization for a reason other than syncope work-up (i.e. unable to cope at home).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator will study the effect of Knowledge Translation on physicians involved in ED syncope care and the effect of the practice recommendations on patients, ED management and safety in 30-days and in 1-year. As the unit of randomization is the ED, all patients presenting to the ED with syncope among whom no serious condition was identified during the index ED evaluation and who did not require consultation/ hospitalization for a non-syncope related reason will be included in the study for analysis. The investigator will use the Canadian Emergency Department Information System presenting complaints suggestive of syncope/pre-syncope or an ED discharge diagnosis of syncope using discharge diagnoses fields or ICD-10 code R.55 for syncope to identify patients.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing the practice recommendations. | The intervention period of 6 months
  To assess the reach of the intervention. We will adopt a pragmatic application of the RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) framework to evaluate the pilot study outcomes. The primary feasibility outcome is the Reach or penetration, the proportion of eligible patients who had the intervention applied.
Rate of hospitalization | At time of ED disposition, an average timeframe is 6 hours
  To assess the impact on hospitalizations.

SECONDARY OUTCOMES:
Rate of consultation | at 6 hours from time of ED disposition
  To assess the effectiveness of intervention on consultation performed in the ED
Mortality | within 30-days and 1-year of the index ED visit
  To assess mortality within 30-days and 1-year of the index ED visit
Rate of adoption | The intervention period of 6 months
  To assess the adoption of CSRS practice recommendation
Number of return ED visits | within 30-days and 1-year
  To assess return ED visits within 30-days and 1-year of the index ED visit
Rate of adherence | The intervention period of 6 months
  To assess the adherence of the CSRS practice recommendation in the ED
Rate of acceptability | The intervention period of 6 months
  To assess the acceptability of the CSRS practice recommendation in the ED
ED disposition time | At time of ED disposition, an average timeframe is 6 hours
  The ED disposition time more accurately reflects the active phase of ED physician care for collecting clinical information, work-up of patients and resolution of diagnostic uncertainty. The longer interval of ED length of stay includes wait times both before and after, which are often determined by triage acuity as well as extraneous system factors (e.g. ED and hospital crowding, staffing patterns, sudden influx of patients, availability of inpatient beds and overcapacity protocols, and availability of transportation for a subgroup patients for whom a decision to discharge has been made).
Degree of satisfaction of the use of CSRS practice recommendation | The intervention period of 6 months
  To assess the satisfaction for the intervention received including support and resources

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandamoorthy, CCFP-EM, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Queensway-Carleton hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Thiruganasambandamoorthy V, Keller M, Nguyen PAI, Gupta P, Ghaedi B, Cao GZQ, Cheung WJ, Khatiwada B, Nemnom MJ, Yadav K, Eagles D, Brehaut J, Tarhuni W, Rouleau G, Desveaux L, Taljaard M. Implementation of the Canadian syncope pathway: a pilot non-randomized stepped wedge trial. CJEM. 2023 Oct;25(10):808-817. doi: 10.1007/s43678-023-00570-7. Epub 2023 Aug 31. PMID 37651075